CLINICAL TRIAL: NCT03113188
Title: Phase 1b Clinical Study of CBP501, Cisplatin and Nivolumab Administered Every 3 Weeks in Patients With Advanced Refractory Tumors
Brief Title: CBP501, Cisplatin and Nivolumab in Advanced Refractory Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CanBas Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBP17-01
Record Dates: First submitted 2017-04-09; First posted 2017-04-13 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2020-10

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Cdc25C phosphatase (211-221)

STUDY DESIGN:
Intervention Model Description: Dose finding cohort plus confirmatory expansion cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CBP501, CDDP, Nivolumab (Experimental): CBP501, Cisplatin and Nivolumab Administered Every 3 Weeks in Patients with Advanced Refractory Tumors
  Interventions: Drug: CBP501

INTERVENTIONS:
Drug: CBP501 — CBP501, CDDP plus Nivolumab

SUMMARY:
This is a multicenter, open-label, phase 1b study of CBP501/cisplatin/nivolumab combination administered once every 21 days to patients with advanced solid tumors.

DETAILED DESCRIPTION:
Multicenter, open-label, phase 1b study of CBP501/cisplatin/nivolumab combination administered once every 21 days to patients with advanced solid tumors. The study will be conducted in two parts.

The first part of the study involves dose-escalation, in which successive cohorts of three patients (expanded up to six patients in the event of a dose-limiting toxicity (DLT) or safety concerns) will receive escalating doses of CBP501 and/or cisplatin until the maximum tolerated dose (MTD) is reached or RP2D defined, based on tolerability observed during the first 21 days of treatment and safety review of all available information by the Safety Monitoring Committee.

The second part of the study involves treatment of expansion cohorts of 10 evaluable patients each in pretreated metastatic exocrine pancreatic cancer and in microsatellite stable colorectal cancer to confirm the tolerability of treatment at the RP2D and evaluate preliminary evidence of anti-tumor activity in these indications.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained prior to initiation of any study-specific procedures and treatment;
2. Previously treated, pathologically confirmed, locally advanced or metastatic solid tumors with measurable disease for which cisplatin is a reasonable treatment option, including, but not limited to, non-small cell lung, mesothelioma, head & neck, ovarian, endometrial, breast, bladder, kidney, esophageal, gastric, colon, liver, gallbladder, cholangiocarcinoma, pancreas, soft tissue sarcoma, and osteosarcoma (for the expansion cohorts, only metastatic exocrine pancreatic cancer and microsatellite stable colorectal cancer are allowed). There is no limit on the number of prior lines of chemotherapy (including prior cisplatin), chemoradiotherapy, radiotherapy or investigational agents the patient can have received in order to be eligible, as long as cisplatin is a reasonable treatment option and all eligibility criteria are met, with the exception that a patient must not have received more than two prior lines incorporating anti-PD-1, anti-PD-L1, or anti-CTLA-4 immune checkpoint blockade.

   Patients who have received prior anti-PD-1, anti-PD-L1, or anti-CTLA-4 immune checkpoint blockade therapy must have tolerated therapy with no evidence of grade 4 toxicity or an immune-related event (any grade) that required treatment discontinuation. Patients who experienced an endocrine related dysfunction are eligible, provided they are on stable hormone replacement therapy;
3. Male or female patients aged ≥ 18 years at time of informed consent;
4. ECOG Performance Status (PS) 0-1;
5. Life expectancy > 3 months;
6. Previous anticancer treatment must be discontinued at least 3 weeks prior to the initiation of study treatment (6 weeks for mitomycin C; 6 weeks for anti-androgen therapy if discontinued prior to treatment initiation, except 8 weeks for bicalutamide);
7. Adequate bone marrow reserve, cardiac, liver, renal and metabolic function:

   * absolute neutrophil count (ANC) ≥ 1.5 x 109/L;
   * platelet count ≥ 100 x 109/L;
   * hemoglobin ≥ 9 g/dL;
   * white blood cell count (WBC) ≤ upper limit of normal (ULN);
   * creatinine phosphokinase isozymes CPK-MB and CPK-MM

     ≤ ULN;
   * serum troponin T levels within normal limits;
   * bilirubin ≤ 1.5 x ULN;
   * alanine aminotransferase (ALT, SGPT) and aspartate aminotransferase (AST, SGOT) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases are present);
   * INR ≤ 1.5 x ULN;
   * serum creatinine ≤ ULN or creatinine clearance ≥ 60 mL/min (by Cockroft & Gault formula or alternate calculation by 24hr urine collection);
   * serum potassium NCI-CTCAE version 4.03 Grade <2;
   * serum calcium NCI-CTCAE version 4.03 Grade <2;
   * serum magnesium NCI-CTCAE version 4.03 Grade <2;
8. Female patients of child-bearing potential must have a negative serum pregnancy test and use at least one form of contraception as approved by the investigator for 4 weeks prior to initiating study treatment and 4 months after the last dose of study drug. For the purposes of this study, child-bearing potential is defined as "all female patients unless they are post-menopausal for at least 3 years or surgically sterile";
9. Male patients must use a form of barrier contraception approved by the investigator during the study and for 4 months after the last dose of study drug;
10. Ability to cooperate with study treatment and follow-up.

Exclusion Criteria

1. Radiation therapy to >30% of bone marrow prior to study entry;
2. Prior chemotherapy with nitrosoureas, prior mitomycin C cumulative dose ≥ 25 mg/m2, prior bone marrow transplant, or prior intensive chemotherapy with stem cell support;
3. Presence of any serious concomitant systemic disorders incompatible with the study in the opinion of the investigator (e.g., uncontrolled congestive heart failure, active infection, etc.);
4. Any previous history of another malignancy (other than cured basal cell or squamous cell carcinoma of the skin or cured in-situ carcinoma) within 5 years of study entry;
5. Presence of any significant central nervous system (CNS) or psychiatric disorder(s) that would hamper the patient's compliance;
6. Evidence of peripheral neuropathy > grade 1 by NCI-CTCAE version 4.03;
7. Treatment with any other investigational agent or participation in another clinical trial within 28 days prior to study entry;
8. Pregnant or breast-feeding patients or any patient with child-bearing potential not using adequate contraception;
9. Known HIV, HBV, or HCV infection (excluding cured HCV infection);
10. Active CNS metastases; however, patients with CNS metastases will be eligible if they have been treated and are stable without symptoms for 4 weeks after completion of treatment, with image documentation required, and must be off steroids;
11. Who require chronic systemic steroid therapy or on any other form of immunosuppressive medication;
12. Has received a live-virus vaccination within 30 days of planned treatment start;
13. With known risk factors for bowel perforation, i.e., history of diverticulitis, intra-abdominal abscess, intestinal obstruction, or abdominal carcinomatosis;
14. Has an active autoimmune disease or a documented history of autoimmune disease;
15. Has a history pneumonitis or interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Recommended dose | 21 days
  Define the recommended doses (RP2D) of CBP501, cisplatin and nivolumab when administered in combination once every 21 days in patients with previously treated advanced solid tumors

SECONDARY OUTCOMES:
Hint of efficacy in pretreated pancreatic and micro-satellite stable colorectal cancer patients | through study completion, an average of 6 month
  Overall response rate will be analyzed according to Simon optimal stage 1 design

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey I Shapiro, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - HonorHealth, Scottsdale, Arizona
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mine N, Yamamoto S, Kufe DW, Von Hoff DD, Kawabe T. Activation of Nrf2 pathways correlates with resistance of NSCLC cell lines to CBP501 in vitro. Mol Cancer Ther. 2014 Sep;13(9):2215-25. doi: 10.1158/1535-7163.MCT-13-0808. Epub 2014 Jul 22. PMID 25053821
- [Background] Krug LM, Wozniak AJ, Kindler HL, Feld R, Koczywas M, Morero JL, Rodriguez CP, Ross HJ, Bauman JE, Orlov SV, Ruckdeschel JC, Mita AC, Fein L, He X, Hall R, Kawabe T, Sharma S. Randomized phase II trial of pemetrexed/cisplatin with or without CBP501 in patients with advanced malignant pleural mesothelioma. Lung Cancer. 2014 Sep;85(3):429-34. doi: 10.1016/j.lungcan.2014.06.008. Epub 2014 Jul 5. PMID 25047675
- [Background] Matsumoto Y, Shindo Y, Takakusagi Y, Takakusagi K, Tsukuda S, Kusayanagi T, Sato H, Kawabe T, Sugawara F, Sakaguchi K. Screening of a library of T7 phage-displayed peptides identifies alphaC helix in 14-3-3 protein as a CBP501-binding site. Bioorg Med Chem. 2011 Dec 1;19(23):7049-56. doi: 10.1016/j.bmc.2011.10.004. Epub 2011 Oct 7. PMID 22032894
- [Background] Mine N, Yamamoto S, Saito N, Yamazaki S, Suda C, Ishigaki M, Kufe DW, Von Hoff DD, Kawabe T. CBP501-calmodulin binding contributes to sensitizing tumor cells to cisplatin and bleomycin. Mol Cancer Ther. 2011 Oct;10(10):1929-38. doi: 10.1158/1535-7163.MCT-10-1139. Epub 2011 Aug 10. PMID 21831962
- [Background] Shapiro GI, Tibes R, Gordon MS, Wong BY, Eder JP, Borad MJ, Mendelson DS, Vogelzang NJ, Bastos BR, Weiss GJ, Fernandez C, Sutherland W, Sato H, Pierceall WE, Weaver D, Slough S, Wasserman E, Kufe DW, Von Hoff D, Kawabe T, Sharma S. Phase I studies of CBP501, a G2 checkpoint abrogator, as monotherapy and in combination with cisplatin in patients with advanced solid tumors. Clin Cancer Res. 2011 May 15;17(10):3431-42. doi: 10.1158/1078-0432.CCR-10-2345. Epub 2011 Jan 10. PMID 21220472
- [Background] Sha SK, Sato T, Kobayashi H, Ishigaki M, Yamamoto S, Sato H, Takada A, Nakajyo S, Mochizuki Y, Friedman JM, Cheng FC, Okura T, Kimura R, Kufe DW, Vonhoff DD, Kawabe T. Cell cycle phenotype-based optimization of G2-abrogating peptides yields CBP501 with a unique mechanism of action at the G2 checkpoint. Mol Cancer Ther. 2007 Jan;6(1):147-53. doi: 10.1158/1535-7163.MCT-06-0371. PMID 17237275